CLINICAL TRIAL: NCT05861076
Title: Moringa Powder Acceptability Trial Among Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022-10-15659
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Consumption; Acceptability; Side Effect

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Baseline assessor will reveal the participants group, only after completing the baseline measurements. After provision of corresponding dosage (assignment), the group information will again be covered, per programming in the Excel file.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moringa Powder - Medium Dose (Experimental): Group A
  Interventions: Other: Moringa Powder - Medium Dose
- Moringa Powder - High Dose (Experimental): Group B
  Interventions: Other: Moringa Powder - High Dose
- Moringa Powder - Low Dose (Experimental): Group C
  Interventions: Other: Moringa Powder - Low Dose

INTERVENTIONS:
Other: Moringa Powder - Low Dose — 1 teaspoon Moringa leaf powder to be consumed with usual food and/or drinks daily for 7 days
  Arms: Moringa Powder - Low Dose
Other: Moringa Powder - Medium Dose — 2 teaspoons Moringa leaf powder to be consumed with usual food and/or drinks daily for 7 days
  Arms: Moringa Powder - Medium Dose
Other: Moringa Powder - High Dose — 3 teaspoons Moringa leaf powder to be consumed with usual food and/or drinks daily for 7 days
  Arms: Moringa Powder - High Dose

SUMMARY:
The study is a randomized acceptability trial involving the provision of three different doses of Moringa powder to be consumed daily by study participants.

DETAILED DESCRIPTION:
Moringa is a drought-resistant nutrient-dense tree with high concentrations of anti-inflammatory plant chemicals in its edible leaves and seeds. In preclinical studies Moringa has been shown to improve insulin resistance, dyslipidemia, and high blood pressure. But its effects in humans remain unclear. Moringa (20g leaf powder on two different days) supplementation decreased post-prandial glucose in Saharawi refugees with type 2 diabetes, compared to controls (Leone, et. al., 2018). In a randomized control trial in Spain, Moringa consumed as six daily capsules of dry leaf powder (2.4 g/day) for 12 weeks, significant decreased fasting blood glucose and glycated hemoglobin (HbA1c) among prediabetic subjects (Gomez-Martinez, et. al., 2021).

The investigators are conducting a testing trial of Moringa oleifera leaves, offered as powder, to be added to foods and/or drinks to test safety, acceptability and consumption of it in three different doses: 1 tsp, 2 tsp, and 3 tsp. Study participants will be randomly allocated to one of the three doses.

Among the studies that have been conducted with human subjects (individuals with diabetes), no adverse effects have been reported with whole leaf powder at up to a single dose of 50 g or using 8 g per day dose for 40 days (Stohs & Hartman, 2015).

The outcomes to be measured in this testing trial are the following:

* Consumption (measured by self-report and skin carotenoid level, as a biomarker of consumption of fruits and vegetables)
* Acceptability (measured by rating the taste of the moringa powder when consumed with foods/drinks)
* Safety (measured by self-report of any potential side effects, such as digestive issues due to fiber content) Results from this trial will suggest an acceptable dose in a population not yet diagnosed with a specific disease (e.g. diabetes) and therefore potentially less willing to consume it in doses that could make taste a potential barrier for consumption.

ELIGIBILITY:
Inclusion Criteria:

* adults (18-65 y old)
* University of California (UC) Berkeley staff
* able to communicate in English or Spanish

Exclusion Criteria:

* UC Berkeley students or academic employees
* pregnant or lactating individuals
* individuals who already consume Moringa regularly
* individuals who have been told that they have diabetes or hypothyroidism
* individuals who are taking any medication, with the exception of over-the-counter pain medication and contraceptives
* individuals who follow a medically prescribed diet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Consumption | 7 days
  Total number of days that moringa powder was consumed
Acceptability | 7 days
  Total acceptability score, in a scale from 3 to 15 points, with higher scores indicating greater acceptance
Side effects | 7 days
  Total number of side effects reported

SECONDARY OUTCOMES:
Daily dose consumed | 7 days
  Average number of teaspoons consumed (among days when consumption was reported)

OTHER OUTCOMES:
Change in skin carotenoids | 7 days
  Difference in skin carotenoid score from baseline to endline (score at endline minus score at baseline). Skin carotenoid levels are measured using the VeggieMeter. This measurement involves scanning a finger using a quick, non-invasive optical method that requires the participant to gently press a finger against a lens surface, with the help of a spring-loaded cover. Skin carotenoids are a biomarker for consumption of fruits and vegetables. A positive outcome value is expected as an indication of consumption of the Moringa powder.
Taste | 7 days
  Average taste score (possible scores range is 1-3, with higher scores indicating greater acceptance)
Texture | 7 days
  Average texture score (possible scores range is 1-3, with higher scores indicating greater acceptance)
Visual appearance | 7 days
  Average visual appearance score (possible scores range is 1-3, with higher scores indicating greater acceptance)
Willingness to continue | 7 days
  Proportion who indicate willingness to continue consuming moringa powder

CONTACTS AND LOCATIONS:
Overall Officials: Susana Matias, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- University of California, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gomez-Martinez S, Diaz-Prieto LE, Vicente Castro I, Jurado C, Iturmendi N, Martin-Ridaura MC, Calle N, Duenas M, Picon MJ, Marcos A, Nova E. Moringa oleifera Leaf Supplementation as a Glycemic Control Strategy in Subjects with Prediabetes. Nutrients. 2021 Dec 24;14(1):57. doi: 10.3390/nu14010057. PMID 35010932
- [Background] Leone A, Bertoli S, Di Lello S, Bassoli A, Ravasenghi S, Borgonovo G, Forlani F, Battezzati A. Effect of Moringa oleifera Leaf Powder on Postprandial Blood Glucose Response: In Vivo Study on Saharawi People Living in Refugee Camps. Nutrients. 2018 Oct 12;10(10):1494. doi: 10.3390/nu10101494. PMID 30322091
- [Background] Stohs SJ, Hartman MJ. Review of the Safety and Efficacy of Moringa oleifera. Phytother Res. 2015 Jun;29(6):796-804. doi: 10.1002/ptr.5325. Epub 2015 Mar 24. PMID 25808883
- See also: Stohs SJ, Hartman MJ. (2015). Review of the Safety and Efficacy of Moringa oleifera. — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC6680322/

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-07-30): https://cdn.clinicaltrials.gov/large-docs/76/NCT05861076/SAP_000.pdf